CLINICAL TRIAL: NCT03974386
Title: Effects of Endotoxin Absorption and Cytokine Removal Hemofilter on Patients With Severe Septic Shock
Brief Title: Effects of Endotoxin Absorption and Cytokine Removal Hemofilter on Severe Septic Shock
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201808098DIPC
Record Dates: First submitted 2019-06-02; First posted 2019-06-04 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Sepsis, Severe; Septic Shock
Keywords: critical care; septic shock; hemofiltration; endotoxin; cytokine storm; prognosis
MeSH Terms: conditions — Sepsis; Shock, Septic; Cytokine Release Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood Purification (Experimental): Patients will receive resuscitation and treatment according to current guidelines for septic shock. In addition to standard care, the patients will receive continuous venovenous hemofiltration and adsorption with oXiris blood purification set.
  Interventions: Device: oXiris blood purification set
- Conventional Treatment (No Intervention): Patients will receive standard care, including resuscitation and treatment according to current guidelines for septic shock.

INTERVENTIONS:
Device: oXiris blood purification set — Continuous venovenous hemofiltration and adsorption (CVVHA) with oXiris filter for up to 72 hours if required. The filter will be replaced every 24 hours. The setting of CVVHA is as follows: blood flow rate 200 mL/min, replacement fluid rate 2000 mL/hr, pre-dilution 50% and post-dilution 50%. If continuous renal replacement therapy is indicated after 72 hours, conventional hemofiltration filters will be used.
  Arms: Blood Purification

SUMMARY:
In recent years, many studies have pointed out that bacterial toxin and cytokine storm are the main causes of shock and multiple organ failure in patients with sepsis. Endotoxin is the main vehicle for systemic inflammatory reaction caused by gram-negative bacteria which induce sepsis. Endotoxin binds to Toll- Like receptor 4 (TLR4) trigger a cytokine storm. The amount of endotoxin is associated with shock, insufficient intestinal perfusion, and poor prognosis. Therefore, clinicians try to use various methods to antagonize the action of endotoxin, which can reduce the cytokine storm and inflammatory response to improve the prognosis of sepsis.

Continuous venous venous hemofiltration plays a role in blood purification in septic shock. With different hemofiltration filters, it has different effects. By removing the inflammatory mediators caused by bacterial toxins and cytokines, shock can be improved. The study plans to receive patients with septic shock and use a hemofiltration filter that adsorbs endotoxin and removes cytokines (oXiris, Baxter Healthcare) to perform continuous venous venous hemofiltration in addition to basic septic shock resuscitation. The effect on the concentration of cytokines in the blood, the infusion dose of inotropics, the fluid balances, and the degree of organ damage was evaluated. It is hoped that the results of this pilot study can lead us to subsequent randomized clinical trials to explore whether this filter can improve the prognosis of septic shock patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet all criteria (A+B+C):
* A) Identified infection source under adequate treatment
* B) Sepsis (the sequential organ failure assessment score rise 2 points or more)
* C) Severe septic shock (serum lactate > 2 mmol/L; need continuous norepinephrine infusion to maintain adequate blood pressure, of which dosage is > 0.2 mcg/kg/min for more than 1 hour or >0.1 mcg/kg/min for more than 3 hours )

Exclusion Criteria:

* Onset of severe septic shock more than 24 hours
* Received continuous renal replacement therapy within 24 hours before enrollment
* Serum white blood cell count count < 1000 cells/μL or Platelet count < 50000 cells/μL
* History of allergy to heparin
* Received cardiopulmonary resuscitation within 4 weeks before enrollment
* ICU admission due to severe septic shock within 2 months
* Patients or Family had chosen palliative care and signed an agreement to deny aggressive treatment
* Pregnancy
* APACHE II Score > 30 at enrollment
* Non-native speakers

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-07-17 (Actual); Study Completion 2020-08-20 (Actual)

PRIMARY OUTCOMES:
Difference of serum interleukin-6 level | 24 hours
  Comparison to enrollment or between 2 groups

SECONDARY OUTCOMES:
Difference of serum interleukin-6 level | 48 hours
  Comparison to enrollment or between 2 groups
Difference of serum interleukin-6 level | 72 hours
  Comparison to enrollment or between 2 groups
Difference of serum interleukin-1β level | 24 hours
  Comparison to enrollment or between 2 groups
Difference of serum interleukin-1β level | 48 hours
  Comparison to enrollment or between 2 groups
Difference of serum interleukin-1β level | 72 hours
  Comparison to enrollment or between 2 groups
Difference of serum interleukin-10 level | 24 hours
  Comparison to enrollment or between 2 groups
Difference of serum interleukin-10 level | 48 hours
  Comparison to enrollment or between 2 groups
Difference of serum interleukin-10 level | 72 hours
  Comparison to enrollment or between 2 groups
Difference of serum procalcitonin level | 24 hours
  Comparison to enrollment or between 2 groups
Difference of serum procalcitonin level | 48 hours
  Comparison to enrollment or between 2 groups
Difference of serum procalcitonin level | 72 hours
  Comparison to enrollment or between 2 groups
Difference of mean arterial pressure | 24 hours
  Comparison to enrollment
Difference of mean arterial pressure | 48 hours
  Comparison to enrollment
Difference of mean arterial pressure | 72 hours
  Comparison to enrollment
Difference of cardiac output | 24 hours
  Comparison to enrollment
Difference of cardiac output | 48 hours
  Comparison to enrollment
Difference of cardiac output | 72 hours
  Comparison to enrollment
Difference of norepinephrine infusion rate | 24 hours
  Comparison to enrollment
Difference of norepinephrine infusion rate | 48 hours
  Comparison to enrollment
Difference of norepinephrine infusion rate | 72 hours
  Comparison to enrollment
Difference of the sequential organ failure assessment score | 24 hours
  Comparison to enrollment or between 2 groups
Difference of the sequential organ failure assessment score | 48 hours
  Comparison to enrollment or between 2 groups
Difference of the sequential organ failure assessment score | 72 hours
  Comparison to enrollment or between 2 groups
Difference of serum endocan level | 24 hours
  Comparison to enrollment or between 2 groups
Difference of serum endocan level | 48 hours
  Comparison to enrollment or between 2 groups
Difference of serum endocan level | 72 hours
  Comparison to enrollment or between 2 groups
Difference of serum diamine oxidase level | 24 hours
  Comparison to enrollment or between 2 groups
Difference of serum diamine oxidase level | 48 hours
  Comparison to enrollment or between 2 groups
Difference of serum diamine oxidase level | 72 hours
  Comparison to enrollment or between 2 groups
Difference of daily IV fluids | 24 hours
  Comparison between 2 groups
Difference of daily IV fluids | 48 hours
  Comparison between 2 groups
Difference of daily IV fluids | 72 hours
  Comparison between 2 groups

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan